CLINICAL TRIAL: NCT05344742
Title: A Multicenter, Open-label, Phase I Dose-escalation and Dose-expansion Study of Mitoxantrone Hydrochloride Liposome Injection Combination Therapy in Chinese Patients With Advanced Solid Tumors
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection Combination Therapy in Chinese Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-027
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitoxantrone Hydrochloride Liposome Injection and Capecitabine (Experimental): Dose-escalation phase: Patients will receive mitoxantrone hydrochloride liposome injection and capecitabine followed by a 3-week DLT observation period. The initial dose of mitoxantrone hydrochloride liposome injection will be set as 18 mg/m^2, and then the dose will be sequentially escalated to 24 mg/m^2 and 30 mg/m^2. The frequency of administration will be once every three weeks. The fixed dose of capecitabine will be set as 1000 mg/m^2, twice daily, from day 1 to day 14. Every 3 weeks will be set as a treatment cycle, and the administration of drugs is planned for 6 cycles.
  Dose-expansion phase: one dose cohort will be selected for dose-expansion to further evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection and capecitabine, and the administration of drugs is planned for 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection; Drug: Capecitabine
- Mitoxantrone Hydrochloride Liposome Injection and albumin-paclitaxel (Experimental): Dose-escalation phase: Patients will receive mitoxantrone hydrochloride liposome injection and albumin-paclitaxel followed by a 3-week DLT observation period. The initial dose of mitoxantrone hydrochloride liposome injection will be set as 18 mg/m^2, and then the dose is sequentially escalated to 24 mg/m^2 and 30 mg/m^2. The frequency of administration will be once every three weeks. The fixed dose of albumin-paclitaxel will be set as 260 mg/m^2, once every three weeks. Every 3 weeks will be set as a treatment cycle, and the administration of drugs is planned for 6 cycles.
  Dose-expansion phase: one dose cohort will be selected for dose-expansion to further evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection and albumin-paclitaxel, and the administration of drugs is planned for 6 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection; Drug: Albumin-paclitaxel

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome injection — Mitoxantrone hydrochloride liposome injection will be administered intravenously once every 3 weeks (a cycle)
Drug: Capecitabine — The fixed dose of oral capecitabine will be administered 1000mg/m^2, twice daily, from day 1 to day 14.
  Arms: Mitoxantrone Hydrochloride Liposome Injection and Capecitabine
Drug: Albumin-paclitaxel — The fixed dose of albumin-paclitaxel will be set as 260 mg/m^2, once every three weeks.
  Arms: Mitoxantrone Hydrochloride Liposome Injection and albumin-paclitaxel

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety, pharmacokinetics (PK) and efficacy of mitoxantrone hydrochloride liposome injection combination therapy in Chinese patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I dose-escalation and dose-expansion study aimed to evaluate the tolerability, safety, pharmacokinetics and efficacy of mitoxantrone hydrochloride liposome injection combination therapy. This study consists of two phases: dose-escalation phase and dose expansion phase.

The dose-escalation phase will be conducted to determine the maximum tolerated dose (MTD) of mitoxantrone hydrochloride liposome injection combination therapy in patients with advanced solid tumors based on a Rolling-6 design. Patients enrolled in this phase will be allocated to two arms A and B. The patients of A arm will receive mitoxantrone hydrochloride liposome injection and capecitabine followed by a 3-week DLT observation period. The patients of B arm will receive mitoxantrone hydrochloride liposome injection and albumin-paclitaxel followed by a 3-week DLT observation period.

After DLT observation, one dose cohort will be selected for dose-expansion to further explore the safety and efficacy of study drug according to the dose-escalation results. In the dose-expansion phase, patients will receive mitoxantrone hydrochloride liposome injection combination therapy every 3 weeks (q3w, a cycle) until disease progression, intolerable toxicity, death, or withdrawal by investigator or patient decision (a maximum of 6 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand and voluntarily participate in this study and sign informed consent;
* Aged 18-65 years, male or female;
* Patients with advanced solid tumors confirmed by histopathology or cytologically and who have failed standard therapy;
* At least one measurable lesion according to RECIST v1.1 at baseline;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* Adverse events（AEs） from the previous treatment have resolved to ≤ Grade 1 based on CTCAE (except for alopecia, hyperpigmentation and the toxicity without safety risk judged by the investigator);
* Adequate organ function defined as:

  * Absolute neutrophil count (ANC) ≥1.5*10^9/L (No Granulocyte Colony Stimulating Factor treatment within 2 weeks prior to the laboratory test);
  * Hemoglobin ≥ 90 g/L (No red blood cell transfusion within 2 weeks prior to the laboratory test);
  * Platelet count ≥ 100*10^9/L (No platelet transfusion within 2 weeks prior to the laboratory test);
  * Creatinine ≤1.5 upper limit of normal (ULN);
  * Total bilirubin ≤1.5 ULN;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3ULN, ≤ 5ULN for patients with liver metastases;
  * Coagulation: prothrombin time (PT) and International Normalization Ratio (INR) ≤1.5ULN；
* Female patients must have a urine or blood human chorionic gonadotropin（HCG） negative test before enrolment (except for menopause and hysterectomy); Patients and their partners must agree to use effective contraceptives measures during the study until 6 months after the end of the last dose.

Exclusion Criteria:

* History of severe allergy to mitoxantrone hydrochloride or liposomal drugs; allergy to capecitabine or any excipients of its components; previous serious and unexpected reaction to fluoropyrimidine or known allergy to fluorouracil; known complete deficiency of dihydropyrimidine dehydrogenase (DPD) activity; allergy to paclitaxel or human albumin;
* Cerebral or meningeal metastases;
* Life expectancy < 3 months;
* Patients with chronic hepatitis B (HBsAg or HBcAb positive with HBV DNA ≥ 2000 IU/mL), chronic hepatitis C (HCV antibody positive with HCV RNA above the lower limit of detection of the study center), or human immunodeficiency virus (HIV) antibody positive;
* Active bacterial, fungal or viral infections that require intravenous infusion treatment within 1 week prior to the first dose;
* Any anticancer treatment within 4 weeks prior to the first dose (e.g., radiotherapy, targeted therapy, immunotherapy, endocrine therapy, etc.); Traditional Chinese medicine or proprietary Chinese medicine with an approved oncology indication within 2 weeks prior to the first dose;
* Enrolled in any other clinical trials within 4 weeks prior to the first dose;
* Patients have undergone major surgery within 3 months prior to the first dose, or have a surgical schedule during the study period;
* Serious thrombosis or thromboembolism as judged by the investigator within 6 months prior to screening;
* History of additional malignant tumor within 3 years, except for locally curable cancer that has been cured, such as basal or squamous cell skin cancer or in situ prostate, cervical or breast cancer;
* Patients with the following cardiac function defects:

  * Long QTc syndrome or QTc interval > 480 ms;
  * Complete left bundle branch block, II-III degree atrioventricular block (except after pacemaker implantation);
  * Severe, uncontrolled arrhythmias requiring pharmacological treatment;
  * History of chronic congestive heart failure, NYHA grade III~IV;
  * Cardiac ejection fraction < 50% within 6 months prior to screening;
  * Severe heart valve disease (regurgitation or stenosis) requiring medical treatment
  * Uncontrollable hypertension (defined as a measured systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under pharmacological control);
  * ECG evidence of myocardial infarction, unstable angina, history of severe pericardial disease, and acute ischemic or severe conduction system abnormalities within 6 months prior to screening;
* Lactating female;
* Significant gastrointestinal disease during screening, which may affect the intake, transportation or absorption of drugs (such as inability to swallow, chronic diarrhoea, intestinal obstruction, etc.);
* Patients who diagnosed with peripheral nerve dysfunction affect their daily life；
* Serious and/or uncontrolled medical condition that, in the judgment of the investigator, may affect the patient's participation in this study (including, but not limited to: diabetes not effectively controlled, kidney disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, substance abuse, neurological disorders, etc.);
* Not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limit toxicity (DLT) | Up to 21 days after the first dose
  Dose limiting toxicity
Treatment-emergent adverse events (TEAEs): | From the initiation of the first dose to 28 days after the last dose
  TEAE is defined as an event that occurs during treatment and does not exist before treatment or worsens compared to before treatment as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetic profile: Cmax | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Peak Plasma Concentration (Cmax)
Objective response rate (ORR) | Throughout the study completion, up to 3 years
  ORR is defined as the proportion of patients who have a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Disease control rate (DCR) | Throughout the study completion, up to 3 years
  DCR is defined as the proportion of patients who have a response of CR/PR or stable disease (SD) as per RECIST 1.1.
Duration of response (DoR) | Throughout the study completion, up to 3 years
  DoR is defined as the time from the first assessment of CR or PR until the date of first occurrence of progressive disease (PD) as per RECIST 1.1 or death from any cause, whichever occurs first
Progression-free survival (PFS) | Throughout the study completion, up to 3 years
  PFS is defined as the time from the date of first dose until the date of first documented PD as per RECIST 1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | Throughout the study completion, up to 3 years
  OS is defined as the time from the date of first dose until the date of death from any cause.
Pharmacokinetic profile: Tmax | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Time to reach maximum concentration (Tmax)
Pharmacokinetic profile: AUC0-t | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-t)
Pharmacokinetic profile: AUC0-∞ | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-∞)
Pharmacokinetic profile: t1/2 | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Half-time (t1/2)
Pharmacokinetic profile: CL | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Clearance (CL)
Pharmacokinetic profile: Vz | Pre-dose and multiple timepoints up to Cycle 4th (each cycle is 21 days)
  Volume of Distribution (Vz)